CLINICAL TRIAL: NCT03188562
Title: Comparison of Diagnostic and Therapeutic Efficacy of Endobronchial/Endoesophageal Ultrasound and Transcervical Extended Mediastinal Lymphadenectomy in Non-Small-Cell Lung Cancer. A Randomised Controlled Trial
Brief Title: Comparison of Diagnostic and Therapeutic Efficacy of EBUS-TBNA/EUS-FNA and TEMLA in Operable NSCLC.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonary Hospital Zakopane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02/2014
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBUS-TBNA, EUS-NA (Experimental): 1. PET/CT
  2. Transbronchial and Transesophageal endoscopic ultrasound-guided needle aspiration ( EBUS-TBNA, EUS-NA)
  Interventions: Other: PET/CT; Procedure: EBUS-TBNA, EUS-NA
- TEMLA (Experimental): 1. PET/CT
  2. Transcervical Extended Mediastinal Lymphadenectomy (TEMLA)
  Interventions: Other: PET/CT; Procedure: TEMLA

INTERVENTIONS:
Other: PET/CT — Positron Emission Tomography (PET/CT)
Procedure: EBUS-TBNA, EUS-NA — Transbronchial and Transesophageal endoscopic ultrasound-guided needle aspiration ( EBUS-TBNA, EUS-NA) Transbronchial ultrasound examination allow to access upper and lower right paratracheal nodes (2R, 4R), subcarinal (7), hilar and interlobar (10, 11), transesophageal ultrasound examination allow to visualize upper and lower left paratracheal nodes (2L, 4L), subaortic (5), para-aortic (6), subcarinal (7), paraesophageal (8), pulmonary ligament (9) nodes. Furthermore EUS allow to localize mediastinal structures including heart, big vessels, main bronchi, vertebral column and diaphragm and can be used in for visualization of tumor infiltration of surrounding structures especially aorta, pulmonary artery or left atrium.
  Arms: EBUS-TBNA, EUS-NA
Procedure: TEMLA — Transcervical Extended Mediastinal Lymphadenectomy (TEMLA) Transcervical Extended Mediastinal Lymphadenectomy (TEMLA) is minimally invasive surgical technique enabling extensive bilateral lymphadenectomy. The procedure starts from 5-8 cm collar incision in the neck, sternum is elevated with a hook connected to a Rochard frame, both laryngeal recurrent nerves and vagus nerves are visualized. During TEMLA all mediastinal nodal stations except for the pulmonary ligament nodes (9) are removed.
  Arms: TEMLA

SUMMARY:
The aim of the study is prospective comparison of diagnostical and therapeutical efficiency between different methods of mediastinal lymph node preoperative staging in Non-Small-Cell Lung Cancer (NSCLC).

Two hundred patients with histologically/cytologically confirmed clinical stage primary I-IIIA NSCLC will be included. The patients must be fit enough to undergo at least pulmonary lobectomy. Computer Tomography (CT) and Positron Emission Tomography (PET/CT) will be performed in all patients. Subsequently, the patients without evidence of dissemination will be randomized to transbronchial and transesophageal endoscopic ultrasound-guided needle aspiration ( EBUS-TBNA, EUS-NA) or Transcervical Extended Mediastinal Lymphadenectomy (TEMLA). The patients with N3 will be referred to definitive oncological treatment, the patients with N2 metastases will be referred to neoadjuvant treatment and the patients without N2/3 metastases will be operated on. The operative procedure will include at least lobectomy with complete lymphadenectomy, with open or video-assisted (VATS) technique. The patients undergoing sublobar resection will be excluded from this study. Final analysis will include comparison of the diagnostic yield and 5-year survival between the EBUS/EUS and the TEMLA arms.

DETAILED DESCRIPTION:
Non-Small-Cell Lung Cancer (NSCLC) is the most common malicious neoplasm characterized by very bad prognosis: 5-year survival rate is only 15%, and the main factors responsible for unfavorable treatment results are late diagnosis, rapid progression of the tumor and high rate of metastasis. The most important issue before selection of the treatment is to establish presence of the metastasis to nodes on the same side of the body (N2) and to lymph nodes on the other side of the mediastinum or a spread to the supraclavicular nodes (N3).

A presence of metastasis to N2 (stage IIIA) is not an absolute contradiction for the surgical treatment but a discovery of N2 is followed by referral of the patients for neoadjuvant or adjuvant treatment depending if N2 are found before or after surgery. Presence of N3 is a contraindication for surgery and an indication for chemo-radiotherapy.

Preoperative techniques of lymph nodes staging includes CT, PET/CT and endoscopy/ultrasound techniques EBUS-TBNA and EUS-NA. Surgical staging techniques include mediastinoscopy, anterior mediastinotomy, VATS, Video-mediastinoscopic lymphadenectomy (VAMLA) and TEMLA.

Endobronchial Ultrasound guided Transbronchial Needle Aspiration (EBUS-TBNA) and Endoscopic Ultrasound guided Needle Aspiration (EUS-NA) are real-time imagining and biopsy techniques used in lung cancer staging. Transbronchial ultrasound examination allow to access upper and lower right paratracheal nodes (2R, 4R), subcarinal (7), hilar and interlobar (10, 11), transesophageal ultrasound examination allow to visualize upper and lower left paratracheal nodes (2L, 4L), subaortic (5), para-aortic (6), subcarinal (7), paraesophageal (8), pulmonary ligament (9) nodes. Furthermore EUS allow to localize mediastinal structures including heart, big vessels, main bronchi, vertebral column and diaphragm and can be used in for visualization of tumor infiltration of surrounding structures especially aorta, pulmonary artery or left atrium.

Transcervical Extended Mediastinal Lymphadenectomy (TEMLA) is minimally invasive surgical technique enabling extensive bilateral lymphadenectomy. The procedure starts from 5-8 cm collar incision in the neck, sternum is elevated with a hook connected to a Rochard frame, both laryngeal recurrent nerves and vagus nerves are visualized. During TEMLA all mediastinal nodal stations except for the pulmonary ligament nodes (9) are removed.

There are many controversions what is the optimal preoperative staging in patients with NSCLC.

It this prospective randomized study we plan to compare preoperative staging with EBUS/EUS with TEMLA in 200 patients.

The patients with histologically or cytologically proven clinical stage I-IIIA NSCLC will be included.

The other inclusion criteria are no previous cancer treatment history, no medical contraindication to operation with at least pulmonary lobectomy, adequate cardiac and pulmonary function.

All patients will undergo CT and PET/CT. The patients without dissemination of cancer will be randomized into the EBUS/EUS and the TEMLA arms. All patients with mediastinal metastasis discovered during staging will be referred to oncological treatment. Patients without mediastinal involvement will be treated with radical surgical treatment (lobectomy or pneumonectomy with lymphadenectomy) with open or video-assisted (VATS) technique. The patients undergoing sublobar resection will be excluded from this study.

Final analysis will include comparison of the diagnostic yield and 5-year survival between the EBUS/EUS and the TEMLA arms. The study is intended to clarify the issue of the optimal preoperative staging and the possible impact of extended bilateral mediastinal lymphadenectomy on the survival of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically or cytologically proven clinical stage I-IIIA NSCLC
* no medical contraindication to operation with at least pulmonary lobectomy
* adequate cardiac and pulmonary function

Exclusion Criteria:

* previous cancer treatment history

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
comparison of the diagnostic yield of EBUS/EUS and TEMLA | 2 weeks after the end of surgery
  after radical surgical treatment (lobectomy or pneumonectomy with lymphadenectomy)

SECONDARY OUTCOMES:
5-year survival between the EBUS/EUS and the TEMLA arms | 5-year
  individual or phone contact with each patient

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Zielinski, PhD, Study Director — Pulmonary Hospital, Zakopane, Poland
Locations (1):
- Pulmonary Hospital, Zakopane, Poland

IPD SHARING:
Plan to Share IPD: Undecided